CLINICAL TRIAL: NCT06909123
Title: A Reduced Dose of Cabergoline for Lactation Inhibition After Second-Trimester Abortion or Pregnancy Loss
Acronym: LISTA3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 80200
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Lactation Suppressed
MeSH Terms: interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cabergoline 1 mg tab (Active Comparator): After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant will be administered cabergoline 1mg orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Cabergoline
- Cabergoline 0.5 mg tab (Experimental): After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant will be administered cabergoline 0.5mg orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — Cabergoline
  Other Names: Dostinex

SUMMARY:
Most patients seeking abortion care or management of pregnancy loss in the second trimester will lactate, which can be physically and emotionally painful. The efficacy of a one-time dose of cabergoline has been previously demonstrated to prevent breast symptoms for these patients. This study seeks to determine if investigators can more precisely manage these patients with a reduced dose appropriate for the physiology of the second trimester, thereby reducing the medication cost and reducing or eliminating the uncomfortable medication side effects.

DETAILED DESCRIPTION:
Most people do not expect breast engorgement following a second-trimester pregnancy loss yet nearly all report bothersome symptoms. Prolactin is the primary hormone responsible for milk production. The dopamine agonist class, including cabergoline, prevents prolactin release, leading to lactation inhibition. Based on dose-finding studies after a full-term birth, a one-time dose of cabergoline 1 mg is offered for lactation inhibition for full-term fetal/neonatal loss or for those with contraindications to breastfeeding.

Recently, our own research found a single dose of cabergoline 1 mg effectively prevents breast symptoms after a second-trimester abortion or stillbirth. However, cabergoline is relatively expensive and associated with side effects such as dizziness, headache, and nausea.

As serum prolactin levels are much lower in the second trimester, it is plausible that a lower dose of cabergoline may still be effective in preventing lactation following a second-trimester loss. Our overarching hypothesis is that a lower dose of cabergoline given after a second-trimester abortion or pregnancy loss will still prevent breast symptoms while also decreasing the frequency and severity of side effects. A lower dose would additionally save money for the healthcare system and patient. For this pilot study, we first plan to test whether a lower dose of cabergoline can reduce serum prolactin levels to physiologic levels.

This is a pilot double-blinded, gestational-age stratified trial of those with fetal demise, stillbirth, or seeking abortion care between 16- and 26-weeks gestation. The investigators will determine if the proportion of participants receiving cabergoline 0.5 mg with normal serum prolactin level on Day 4 is non-inferior to those receiving cabergoline 1 mg.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people, ages 18 years or older
* Intrauterine pregnancy between 16/0-25/6 weeks of gestation age (by ultrasound dating performed prior to or same day of enrollment visit)
* Consented for an induced, elective abortion or undergoing management of fetal demise
* English or Spanish speaking
* Able to consent for a research study, literate in English or Spanish
* Willing to comply with study procedures and follow-up
* Access to smart phone throughout study

Exclusion Criteria:

* Prior mastectomy (breast reduction or chest masculinization surgery acceptable)
* Currently breastfeeding
* Currently receiving dopamine agonist or antagonist therapy for other indication leg syndrome)
* Contraindication to cabergoline (as per package insert)
* Uncontrolled hypertension - defined as baseline BP > 160/110, or chronic hypertension requiring more than one baseline medication, or current pregnancy-induced hypertension spectrum disorders (gestational hypertension, preeclampsia, eclampsia)
* History of cardiac valvular disorders or valvular repair
* History of pulmonary, pericardial, or retroperitoneal fibrotic disorders

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serum prolactin level less than 23 ng/mL | Day 4
  Comparison of the proportion of participants receiving cabergoline 0.5 mg with normal serum prolactin level (defined as less than 23ng/mL) to those receiving cabergoline 1 mg

SECONDARY OUTCOMES:
Number of participants with breast symptoms | Day 4
  Participants will assess their breast symptoms using the validated Bristol Breast Inventory survey to assess 4 domains of breast symptoms: tenderness, engorgement, leaking milk, pain relief. Participants who indicated symptoms in any of these areas met the criteria for this outcome.

IPD SHARING:
Plan to Share IPD: No